CLINICAL TRIAL: NCT00310076
Title: Phase II Trial of Adjuvant Thalidomide Following Cytoreductive Surgery and Intraperitoneal Hyperthermic Chemotherapy for Peritoneal Carcinomatosis or Adenomucinosis From Colorectal/Appendiceal Cancer
Brief Title: Thalidomide in Treating Patients Who Have Undergone Surgery and Chemotherapy for Cancer That Has Spread Throughout the Abdomen Due to Colorectal Cancer or Appendix Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466311; CCCWFU-59202; CCCWFU-BG02-406; CELGENE-CCCWFU-59202
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma of the Appendix; Colorectal Cancer
Keywords: carcinoma of the appendix; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent colon cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Thalidomide; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemo therapy followed by thalidomide (Experimental): After cytoreductive surgery with intraperitoneal hyperthermic chemotherapy, patients will receive thalidomide orally each evening for 24 months or until tumor progression is detected.
  Interventions: Drug: thalidomide; Procedure: surgery

INTERVENTIONS:
Drug: thalidomide — Patients will receive thalidomide orally each evening for 24 months or until tumor progression is detected.
Procedure: surgery — Cytoreductive Surgery with Intraperitoneal Hyperthermic Chemotherapy

SUMMARY:
RATIONALE: Thalidomide may stop the growth of tumor cells by blocking blood flow to the tumor. Giving thalidomide after surgery and chemotherapy may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well thalidomide works in treating patients who have undergone surgery and received chemotherapy directly into the abdomen by hyperthermic perfusion for cancer that has spread throughout the abdomen due to colorectal cancer or appendix cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine time to progression from surgery in patients who have undergone cytoreductive surgery and intraperitoneal hyperthermic chemotherapy for peritoneal carcinomatosis or adenomucinosis secondary to colorectal or appendiceal cancer treated with adjuvant thalidomide.

Secondary

* Estimate progression-free survival probability of patients treated with this regimen.
* Obtain toxicity data for patients receiving long-term oral thalidomide therapy.

OUTLINE: Patients receive oral thalidomide once daily on days 1-28. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed peritoneal carcinomatosis or adenomucinosis secondary to colorectal or appendiceal cancer

  * Underwent cytoreductive surgery and intraperitoneal hyperthermic chemotherapy (IPHC) within the past 12 weeks

    * Patients with residual disease or no evidence of disease after IPHC are eligible
* No extra-abdominal disease or parenchymal liver metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Free of infection or postoperative complications
* Hemoglobin > 8.0 g/dL
* Absolute neutrophil count > 1,000/mm³
* Platelet count > 100,000/mm³
* PTT or PT < 1.5 times normal (except in patients who are receiving therapeutic anticoagulant therapy for non-related medical conditions, such as atrial fibrillation)
* Bilirubin < 1.5 mg/dL OR direct bilirubin ≤ 1.0 mg/dL (for patients with Gilbert's syndrome)
* AST/ALT ≤ 2.5 times normal
* Serum creatinine < 2.0 mg/dL
* No peripheral neuropathy > grade 1, except localized neuropathy due to a mechanical cause or trauma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception for 4 months prior to, during, and for 4 months after treatment with thalidomide
* No history of hepatic cirrhosis
* No history of severe hypothyroidism
* No history of medical problem such as severe congestive heart failure or active ischemic heart disease
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No known history of deep vein thrombosis or pulmonary embolus

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy, biologic therapy, or radiotherapy (except for IPHC)
* No other concurrent systemic therapy
* No concurrent high level sedatives
* No concurrent sedating "recreational" drugs or alcohol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-10; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Shen, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemo Therapy Followed by Thalidomide
Started | 29
Completed | 26
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chemo Therapy Followed by Thalidomide
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression after surgery was recorded.
Time Frame: 9 hours
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Chemo Therapy Followed by Thalidomide
Number analyzed (Participants) | 26
years | 0.775 [0.42 to 3.38]

2. Secondary Outcome: Progression Free Survival
Time Frame: 60 months after treatment
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Chemo Therapy Followed by Thalidomide
Number analyzed (Participants) | 26
years | 0.775 [0.42 to 3.38]

3. Secondary Outcome: Number of Events of Toxicity Graded 3 and 4
Description: Adverse events with Common Toxicity Criteria grades of 3 and 4 are reported
Time Frame: up to 60 months
Measure: Number; unit: number of events
Arm/Group | Chemo Therapy Followed by Thalidomide
Number analyzed (Participants) | 26
number of events
  Grade 3 | 17
  Grade 4 | 4

ADVERSE EVENTS:
Time Frame: up to 60 months
Arm/Group | Chemo Therapy Followed by Thalidomide
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Therapy Followed by Thalidomide (N=27)
Cardiac Dysrhythmias (Cardiac disorders) | 1 (1)
Cardiovascular/General-other (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia, esophagitis, odynophagia (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
other gastrointestinal (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hypertension (General disorders) | 1 (1)
Hypokalemia (Investigations) | 2 (2)
Hypomagnesemia (Investigations) | 1 (1)
Hypotension (General disorders) | 1 (1)
Hypoxia (General disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 3 (3)
Infection/Febrile Neutropenia-Other (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neuro-mood (Psychiatric disorders) | 2 (2)
Neuro-motor (Psychiatric disorders) | 2 (2)
Neurosensory (Nervous system disorders) | 5 (5)
Pain-other (Nervous system disorders) | 2 (2)
Thrombosis/Embolism (Cardiac disorders) | 2 (2)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight Gain (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Therapy Followed by Thalidomide (N=27)
Leukocytes (Investigations) | 10 (10)
Anorexia (General disorders) | 3 (3)
Alk Phos (Investigations) | 8 (8)
Alopecia (General disorders) | 5 (5)
Edema (Metabolism and nutrition disorders) | 3 (3)
Absolute Neutrophil Count (Investigations) | 3 (3)
Dizziness/vertigo (General disorders) | 4 (4)
Insomnia (General disorders) | 2 (2)
Neurologic Other (Nervous system disorders) | 9 (9)
Dermatological (Skin and subcutaneous tissue disorders) | 7 (7)
Weight Loss (General disorders) | 4 (4)
Hyperglycemia (Investigations) | 14 (14)
Hypoglycemia (Investigations) | 2 (2)
Hypocalcemia (Investigations) | 8 (8)
Hyponatremia (Investigations) | 2 (2)
Coagulation Other (Investigations) | 2 (2)
Hot flashes/flushes (General disorders) | 2 (2)
Endocrine Other (Endocrine disorders) | 3 (3)
Hypoalbuminemia (Investigations) | 4 (4)
Serum glutamic pyruvic transaminase (Investigations) | 7 (7)
Somnolence (General disorders) | 5 (5)
Serum glutamic oxaloacetic transaminase (Investigations) | 5 (5)
Hyperkalemia (Investigations) | 4 (4)
Hypernatremia (Investigations) | 3 (3)
Fever in the absence of neutropenia (Investigations) | 2 (2)
Infection-Other (Infections and infestations) | 2 (2)
Auditory/Ear-Other (Ear and labyrinth disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes